CLINICAL TRIAL: NCT05256303
Title: Hospital-Level Care at Home for Acutely Ill Adults in Rural Settings: A Randomized Controlled Trial
Brief Title: Rural Hospital-Level Care at Home for Acutely Ill Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: The Thompson Family Foundation Inc (Unknown)
Responsible Party: Principal Investigator, David Levine, Dr. David Levine MD, MPH, MA, Director, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2021P000334
Record Dates: First submitted 2021-10-25; First posted 2022-02-25 (Actual); Last update posted 2025-11-12 (Actual); Status verified 2025-11

CONDITIONS: Infections; Heart Failure; Chronic Obstructive Pulmonary Disease; Asthma; Gout Flare; Chronic Kidney Diseases; Hypertensive Urgency; Atrial Fibrillation Rapid; Anticoagulation; Diabetes and Its Complications; End of Life/Desires Only Medical Management
Keywords: home hospital; hospital at home; hospital in the home
MeSH Terms: conditions — Infections; Heart Failure; Pulmonary Disease, Chronic Obstructive; Asthma; Renal Insufficiency, Chronic; Hypertensive Crisis; Diabetes Mellitus | interventions — Home Care Services, Hospital-Based

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Home Hospital care (Experimental): Patients receive hospital-level care in their home, as a substitute to traditional hospital care.
  Interventions: Other: Home Hospital care
- Traditional Hospital care (Active Comparator): Patients receive hospital-level care in the hospital.
  Interventions: Other: Traditional Hospital care

INTERVENTIONS:
Other: Home Hospital care — Patients receive hospital-level care in their home
  Arms: Home Hospital care
Other: Traditional Hospital care — Patients receive hospital-level care in the hospital.
  Arms: Traditional Hospital care

SUMMARY:
This study examines the implications of providing hospital-level care in rural homes.

DETAILED DESCRIPTION:
Home hospital is hospital-level care at home for acutely ill patients. In multiple publications mostly in urban environments, home hospital care delivered cost-effective, high-quality, excellent experience care with similar quality and safety as traditional hospital care. Most home hospital models deliver care in urban environments, not in rural environments.

To determine the effect of home hospital care in rural homes, the investigators propose to the following randomized control trial.

ELIGIBILITY:
Inclusion Criteria:

Patient clinical inclusion criteria:

* >=18 years old
* Any infectious process (e.g., pneumonia, diverticulitis, cellulitis, complicated urinary tract infection)
* Heart failure exacerbation
* Asthma and chronic obstructive pulmonary disease exacerbation
* Atrial fibrillation with rapid ventricular response
* Diabetes and its complications
* Venous thromboembolism
* Gout exacerbation
* Chronic kidney disease with volume overload
* Hypertensive urgency
* End of life / desires only medical management

Patient environmental inclusion criteria:

* Lives in a rural area that can be served by the RHH team.
* Has capacity to consent to study OR can assent to study and has proxy who can consent (see subject enrollment, below)
* Can identify a potential caregiver who agrees to stay with patient for first 24 hours of admission. Caregiver must be competent to call care team if a problem is evident to her/him. After 24 hours, this caregiver should be available for as-needed spot checks on the patient.

  * This criterion may be waived for highly competent patients at the patient and clinician's discretion.

Patient caregiver inclusion criteria: (not required for patient participation):

* Age >= 18 years old
* Has capacity to consent to study
* Lives within 15 minutes travel time.

Clinician inclusion criteria:

* The rural home hospital clinical team will be identified by the site PI at each study site prior to the start of the study. The site PI will recruit local RNs and/or EMT-Ps, and attending physicians (MD) to deploy and provide rural home hospital care.
* Any member of the rural home hospital clinical team (a clinician providing care in the home) who will be participating in research activities, including the screening and recruitment of patients for the rural home hospital intervention and/or providing care to rural patients that enroll in the intervention.

Sites without continuous monitoring will make amendments to the above inclusion criteria

Exclusion Criteria:

* Patient exclusion clinical criteria:

  * Acute delirium, as determined by the Confusion Assessment Method
  * Cannot establish peripheral access by any means
  * Secondary condition: active non-melanoma/prostate cancer, end-stage renal disease, acute myocardial infarction, acute cerebral vascular accident, acute hemorrhage (unless part of end of life pathway)
  * Primary diagnosis requires multiple or routine administrations of intravenous narcotics for pain control
  * Cannot independently ambulate to bedside commode, unless home-based aides are available
  * As deemed by on-call MD, patient likely to require any of the following procedures that have not already occurred: computed tomography, magnetic resonance imaging, endoscopic procedure, blood transfusion, cardiac stress test, or surgery (unless these can be coordinated with appropriate facilities during the home hospitalization)
  * For pneumonia:

    * Most recent CURB65 > 3: new confusion, BUN > 19mg/dL, respiratory rate>=30/min, systolic blood pressure<90mmHg, Age>=65 (<14% 30-day mortality)15
    * Most recent SMRTCO > 2: systolic blood pressure < 90mmHg (2pts), multilobar CXR involvement (1pt), respiratory rate >= 30/min, heart rate >= 125, new confusion, oxygen saturation <= 90% (<10% chance of intensive respiratory or vasopressor support)16
    * Absence of clear infiltrate on imaging
    * Cavitary lesion on imaging
    * Pulmonary effusion of unknown etiology
    * O2 saturation < 90% despite 5L O2
  * For heart failure:

    * Has a left ventricular assist device
    * GWTG-HF17 (>10% in-hospital mortality) or ADHERE18 (high risk or intermediate risk 1)*
    * Severe pulmonary hypertension
  * For complicated urinary tract infection:

    * Absence of pyuria
    * Most recent qSOFA > 1 (SBP≤100 mmHg, RR≥22, GCS<15 [any AMS]) (if sepsis, >10% mortality)19
  * For other infection

    * Most recent qSOFA > 1 (SBP≤100 mmHg, RR≥22, GCS<15 [any AMS]) (if sepsis, >10% mortality)19
  * For COPD

    * BAP-65 score > 3 (BUN>25, altered mental status, HR>109, age>65) (<13% chance in-hospital mortality): exercise caution
  * For asthma

    o Peak expiratory flow < 50% of normal: exercise caution
  * For diabetes and its complications

    o Requires IV insulin
  * For hypertensive urgency

    * Systolic blood pressure > 190 mmHg
    * Evidence of end-organ damage; for example, acute kidney injury, focal neurologic deficits, myocardial infarction
  * For atrial fibrillation with rapid ventricular response

    * Likely to require cardioversion
    * New atrial fibrillation with rapid ventricular response
    * Unstable blood pressure, respiratory rate, or oxygenation
    * Despite IV beta and/or calcium channel blockade in the emergency department, HR remains > 125 and SBP remains different than baseline
    * Less than 1 hour of time has elapsed with HR < 125 and SBP similar or higher than baseline
  * Home hospital census is full

    * GWTG-HF: AHA Get with the Guidelines: SBP, BUN, Na, Age, HR, Black race, COPD ADHERE: Acute decompensated heart failure national registry: BUN, creatinine, SBP

Patient environmental exclusion criteria:

* Undomiciled
* No working heat (October-April), no working air conditioning if forecast > 80°F (June-September), or no running water
* On methadone requiring daily pickup of medication
* In police custody
* Resides in facility that provides on-site medical care (e.g., skilled nursing facility)
* Domestic violence screen positive

Sites without continuous monitoring will make amendments to the above exclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2022-02-16 (Actual); Primary Completion 2023-12-17 (Actual); Study Completion 2024-01-17 (Actual)

PRIMARY OUTCOMES:
Total cost, hospitalization | Date of admission to date of discharge, estimated 10 days later
  Published as percent change given sensitivity of these data

SECONDARY OUTCOMES:
Total cost, discharge to 30-days post discharge | Day of discharge to 30 days later
  Published as percent change given sensitivity of these data
Unplanned readmission within 30-days of discharge | Day of discharge to 30 days later
  Percentage
Days at home | Day of discharge to 30 days later
  The number of days spent at home from the day of discharge to 30-days later
Percent of day lying down | Day of admission to day of discharge, assessed up to 2 months

OTHER OUTCOMES:
Length of stay, days | Day of admission to day of discharge, assessed up to 2 months
  Exploratory
IV medication, days | Day of admission to day of discharge, assessed up to 2 months
  Exploratory
Intravenous fluids, days | Day of admission to day of discharge, assessed up to 2 months
  Exploratory
Intravenous diuretics, days | Day of admission to day of discharge, assessed up to 2 months
  Exploratory
Intravenous antibiotics, days | Day of admission to day of discharge, assessed up to 2 months
  Exploratory
Oxygen requirement, days | Day of admission to day of discharge, assessed up to 2 months
  Exploratory
Nebulizer treatment, days | Day of admission to day of discharge, assessed up to 2 months
  Exploratory
Imaging, % | Day of admission to day of discharge, assessed up to 2 months
  Exploratory
Lab orders, # | Day of admission to day of discharge, assessed up to 2 months
  Exploratory
MD sessions, # of notes | Day of admission to day of discharge, assessed up to 2 months
  Exploratory
Consultant sessions, # of notes | Day of admission to day of discharge, assessed up to 2 months
  Exploratory
PT/OT sessions, # of notes | Day of admission to day of discharge, assessed up to 2 months
  Exploratory
Frequency of disposition, routine, SNF, home health, other | Day of admission to day of discharge, assessed up to 2 months
  Exploratory
Follow up with patient's PCP within 14 days, y/n | Up to 30 days from day of discharge, assessed up to 2 months
  Exploratory
SNF utilization, days | Up to 30 days from day of discharge, assessed up to 2 months
  Exploratory
Home health utilization, days | Up to 30 days from day of discharge, assessed up to 2 months
  Exploratory
Unplanned readmission(s) after index, # and y/n + date | Up to 30 days from day of discharge, assessed up to 2 months
  Exploratory
ED observation stay(s), # and y/n + date | Up to 30 days from day of discharge, assessed up to 2 months
  Exploratory
ED visit(s), # and y/n + date | Up to 30 days from day of discharge, assessed up to 2 months
  Exploratory
Fall, y/n | Day of admission to day of discharge, assessed up to 2 months
  Exploratory
Delirium, y/n | Day of admission to day of discharge, assessed up to 2 months
  Exploratory
DVT/PE, y/n | Day of admission to day of discharge, assessed up to 2 months
  Exploratory
New pressure ulcer, y/n | Day of admission to day of discharge, assessed up to 2 months
  Exploratory
Thrombophlebitis at peripheral IV site, y/n | Day of admission to day of discharge, assessed up to 2 months
  Exploratory
Hospital-acquired catheter-associated urinary tract infection, y/n | Day of admission to day of discharge, assessed up to 2 months
  Exploratory
Hospital-acquired Clostridium difficile infection, y/n | Day of admission to day of discharge, assessed up to 2 months
  Exploratory
Hospital-acquired methicillin resistant staphylococcus aureus infection, y/n | Day of admission to day of discharge, assessed up to 2 months
  Exploratory
New arrhythmia, y/n | Day of admission to day of discharge, assessed up to 2 months
  Exploratory
Hypokalemia, y/n | Day of admission to day of discharge, assessed up to 2 months
  Exploratory
Acute kidney injury, y/n | Day of admission to day of discharge, assessed up to 2 months
  Exploratory
Medication error, y/n | Day of admission to day of discharge, assessed up to 2 months
  Exploratory
Unanticipated mortality, y/n | Day of admission to day of discharge, assessed up to 2 months
  Exploratory
Loss of consciousness, y/n | Day of admission to day of discharge, assessed up to 2 months
  Exploratory
Transfer back to hospital, y/n | Day of admission to day of discharge, assessed up to 2 months
  Intervention arm only; Exploratory
Unplanned mortality during admission | Day of admission to day of discharge, assessed up to 2 months
  Exploratory
Unplanned 30-day mortality | Day of discharge to 30-days post discharge, assessed up to 2 months
  Exploratory
Pain management, mean pain score on a scale from 0-10 where 10 is the worst pain imaginable | Day of admission to day of discharge, assessed up to 2 months
  Exploratory
Hours of sleep per day | Day of admission to day of discharge, assessed up to 2 months
  Exploratory
Hours of sleep per night | Day of admission to day of discharge, assessed up to 2 months
  Exploratory
Hours of activity per day | Day of admission to day of discharge, assessed up to 2 months
  Exploratory
Hours of activity per night | Day of admission to day of discharge, assessed up to 2 months
  Exploratory
Hours of sitting upright per day | Day of admission to day of discharge, assessed up to 2 months
  Exploratory
Hours of sitting upright per night | Day of admission to day of discharge, assessed up to 2 months
  Exploratory
Daily steps | Day of admission to day of discharge, assessed up to 2 months
  Exploratory
Use of inappropriate medications in the elderly, y/n | Day of admission to day of discharge, assessed up to 2 months
  Exploratory
Use of Foley catheter, y/n | Day of admission to day of discharge, assessed up to 2 months
  Exploratory
Use of restraints, y/n | Day of admission to day of discharge, assessed up to 2 months
  Exploratory
EuroQol-5D-5L, visual analogue scale, 0-100, where 100 is the best imaginable health today | At admission, at discharge (the day the patient leaves the hospital environment), and at 30 days after discharge, each assessed up to 2 months
  Exploratory
SF-1 | At admission, at discharge (the day the patient leaves the hospital environment), and at 30 days after discharge, each assessed up to 2 months
  Exploratory; 1-5 Likert scale: Excellent, very good, good, fair poor
Activities of daily living, score | At admission, at discharge (the day the patient leaves the hospital environment), and at 30 days after discharge, each assessed up to 2 months
  Exploratory
Instrumental activities of daily living, score | At admission, at discharge (the day the patient leaves the hospital environment), and at 30 days after discharge, each assessed up to 2 months
  Exploratory
Patient health questionnaire-2, score | At admission, at discharge (the day the patient leaves the hospital environment), and at 30 days after discharge, each assessed up to 2 months
  Exploratory
PROMIS Emotional Support Short Form 4a, score | At admission, at discharge (the day the patient leaves the hospital environment), and at 30 days after discharge, each assessed up to 2 months
  Exploratory; I have someone who will listen to me when I need to talk I have someone to confide in or talk to about myself or my problems I have someone who makes me feel appreciated I have someone to talk with when I have a bad day Scale for each: never, rarely, sometimes, usually, always
Picker Experience Questionnaire -15, score, measured 0-15, where 15 is the best patient experience | Within 30 days after discharge, assessed up to 2 months
  Exploratory
Global satisfaction with care, score, 0-10, where 10 is the best global satisfaction | Within 30 days after discharge, assessed up to 2 months
  Exploratory
Recommend care, score, 0-10, where 10 is the best recommendation possible | Within 30 days after discharge, assessed up to 2 months
  Exploratory
Qualitative interview | Day of discharge to 30 days after discharge, assessed up to 2 months
  Exploratory
Caregiver burden (Zarit), 0-48, where 48 indicates the worst possible caregiver burden | Day of admission and within 30 days after discharge, assessed up to 2 months
  Exploratory
Number of RN visits, in-person | Day of admission to day of discharge, assessed up to 2 months
  Exploratory
Number of RN visits, virtual | Day of admission to day of discharge, assessed up to 2 months
  Exploratory
Number of RN visits, total | Day of admission to day of discharge, assessed up to 2 months
  Exploratory
RN travel time | Day of admission to day of discharge, assessed up to 2 months
  Exploratory
Failed connectivity, % | Day of admission to day of discharge, assessed up to 2 months
  Exploratory
Number of "on call" MD interactions (video or phone) | Day of admission to day of discharge, assessed up to 2 months
  Exploratory
Duration of 1st RN visit | Day of admission, assessed up to 2 months
  Exploratory
Duration of subsequent RN visit, in-person | Day of admission to day of discharge, assessed up to 2 months
  Exploratory
Duration of subsequent RN visit, virtual | Day of admission to day of discharge, assessed up to 2 months
  Exploratory
Other metrics captured on the clinician process survey and nursing visit form | Day of admission to day of discharge, assessed up to 2 months
  Exploratory
Insufficient handoff | Day of admission to day of discharge, assessed up to 2 months
  Exploratory
Documentation error | Day of admission to day of discharge, assessed up to 2 months
  Exploratory
Equipment malfunction | Day of admission to day of discharge, assessed up to 2 months
  Exploratory
Age | Day of admission, assessed up to 2 months
  Exploratory
Gender | Day of admission, assessed up to 2 months
  Exploratory
Race/ethnicity | Day of admission, assessed up to 2 months
  Exploratory
Primary language | Day of admission, assessed up to 2 months
  Exploratory
Health insurance states, public/private/none | Day of admission, assessed up to 2 months
  Exploratory
BMI | Day of admission, assessed up to 2 months
  Exploratory
Comorbidities, type and # | Day of admission, assessed up to 2 months
  Exploratory
Partner status | Day of admission, assessed up to 2 months
  Exploratory
Education | Day of admission, assessed up to 2 months
  Exploratory
Zip code | Day of admission, assessed up to 2 months
  Exploratory
Employment | Day of admission, assessed up to 2 months
  Exploratory
Smoking status | Day of admission, assessed up to 2 months
  Exploratory
Medications used as outpatient, # | Day of admission, assessed up to 2 months
  Exploratory
DNR/I code status | Day of admission, assessed up to 2 months
  Exploratory
Lives alone | Day of admission, assessed up to 2 months
  Exploratory
Home health aide prior to admission | Day of admission, assessed up to 2 months
  Exploratory
Elective and urgent admissions in the previous year, # | Day of admission, assessed up to 2 months
  Exploratory
ED visits in the previous 6 months, # | Day of admission, assessed up to 2 months
  Exploratory
Interqual disease-specific leveling | Day of admission, assessed up to 2 months
  Exploratory
PRISMA-7 | Day of admission, assessed up to 2 months
  Exploratory
Eight-item Interview to Differentiate Aging and Dementia | Day of admission, assessed up to 2 months
  Exploratory
Would you be surprised if this patient died in the next year? | Day of admission, assessed up to 2 months
  Exploratory
BRIEF health literacy screening tool | Day of admission, assessed up to 2 months
  Exploratory
Readmission risk score on discharge (HOSPITAL) | Day of discharge, assessed up to 2 months
  Exploratory
Admitting diagnosis | Day of admission, assessed up to 2 months
  Exploratory
Admission source | Day of admission, assessed up to 2 months
  Exploratory
COVID case count on day of admission | Day of admission, assessed up to 2 months
  Exploratory
Degree of rurality | Day of admission, assessed up to 2 months
  Exploratory
[intervention arm only] RHH admission, daily care, and discharge processes accomplished | Twice a week, day of enrollment to day of final discharge, assessed up to 2 months
  Exploratory
[intervention arm only] Perceived acceptability of RHH care | Day of discharge to 30 days postdischarge, assessed up to 2 months
  Exploratory
[intervention arm only] Perceived safety, quality of care, caregiver burden | Day of discharge to 30 days, assessed up to 2 months
  Exploratory
Qualitative interviews | Day of enrollment to day of final discharge, assessed up to 4 months
  Interviews with patients, caregivers, and rural home hospital clinicians.

CONTACTS AND LOCATIONS:
Locations (3):
- United States (2):
  - Blessing Health System, Quincy, Illinois
  - Appalachian Regional Healthcare, Inc., Hazard, Kentucky
- Wetaskiwin Hospital and Care Centre, Wetaskiwin, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hung WW, Ross JS, Farber J, Siu AL. Evaluation of the Mobile Acute Care of the Elderly (MACE) service. JAMA Intern Med. 2013 Jun 10;173(11):990-6. doi: 10.1001/jamainternmed.2013.478. PMID 23608775
- [Background] Fong TG, Tulebaev SR, Inouye SK. Delirium in elderly adults: diagnosis, prevention and treatment. Nat Rev Neurol. 2009 Apr;5(4):210-20. doi: 10.1038/nrneurol.2009.24. PMID 19347026
- [Background] 2014 National and State Healthcare-Associated Infections Progress Report.; 2016. http://www.cdc.gov/hai/surveillance/progress-report/index.html. Accessed April 19, 2016.
- [Background] Counsell SR, Holder CM, Liebenauer LL, Palmer RM, Fortinsky RH, Kresevic DM, Quinn LM, Allen KR, Covinsky KE, Landefeld CS. Effects of a multicomponent intervention on functional outcomes and process of care in hospitalized older patients: a randomized controlled trial of Acute Care for Elders (ACE) in a community hospital. J Am Geriatr Soc. 2000 Dec;48(12):1572-81. doi: 10.1111/j.1532-5415.2000.tb03866.x. PMID 11129745
- [Background] Leff B, Burton L, Mader SL, Naughton B, Burl J, Inouye SK, Greenough WB 3rd, Guido S, Langston C, Frick KD, Steinwachs D, Burton JR. Hospital at home: feasibility and outcomes of a program to provide hospital-level care at home for acutely ill older patients. Ann Intern Med. 2005 Dec 6;143(11):798-808. doi: 10.7326/0003-4819-143-11-200512060-00008. PMID 16330791
- [Background] Cryer L, Shannon SB, Van Amsterdam M, Leff B. Costs for 'hospital at home' patients were 19 percent lower, with equal or better outcomes compared to similar inpatients. Health Aff (Millwood). 2012 Jun;31(6):1237-43. doi: 10.1377/hlthaff.2011.1132. PMID 22665835
- [Background] Levine DM, Ouchi K, Blanchfield B, Diamond K, Licurse A, Pu CT, Schnipper JL. Hospital-Level Care at Home for Acutely Ill Adults: a Pilot Randomized Controlled Trial. J Gen Intern Med. 2018 May;33(5):729-736. doi: 10.1007/s11606-018-4307-z. Epub 2018 Feb 6. PMID 29411238
- [Background] Levine DM, Ouchi K, Blanchfield B, Saenz A, Burke K, Paz M, Diamond K, Pu CT, Schnipper JL. Hospital-Level Care at Home for Acutely Ill Adults: A Randomized Controlled Trial. Ann Intern Med. 2020 Jan 21;172(2):77-85. doi: 10.7326/M19-0600. Epub 2019 Dec 17. PMID 31842232
- [Background] Bureau UC. What is Rural America?https://www.census.gov/library/stories/2017/08/rural-america.html. Published 2017. Accessed May 31, 2019.
- [Background] Garcia MC, Rossen LM, Bastian B, Faul M, Dowling NF, Thomas CC, Schieb L, Hong Y, Yoon PW, Iademarco MF. Potentially Excess Deaths from the Five Leading Causes of Death in Metropolitan and Nonmetropolitan Counties - United States, 2010-2017. MMWR Surveill Summ. 2019 Nov 8;68(10):1-11. doi: 10.15585/mmwr.ss6810a1. PMID 31697657
- [Background] Parker K, Horowitz J, Brown A, Fry R, Cohn D, Igielnik R. What Unites and Divides Urban, Suburban and Rural Communities.; 2018. https://www.pewsocialtrends.org/wpcontent/uploads/sites/3/2018/05/Pew-Research-Center-Community-Type-Full-Report-FINAL.pdf. Accessed May 31, 2019
- [Background] Creditor MC. Hazards of hospitalization of the elderly. Ann Intern Med. 1993 Feb 1;118(3):219-23. doi: 10.7326/0003-4819-118-3-199302010-00011. PMID 8417639
- [Background] Joynt KE, Orav EJ, Jha AK. Mortality rates for Medicare beneficiaries admitted to critical access and non-critical access hospitals, 2002-2010. JAMA. 2013 Apr 3;309(13):1379-87. doi: 10.1001/jama.2013.2366. PMID 23549583
- [Background] Joynt KE, Harris Y, Orav EJ, Jha AK. Quality of care and patient outcomes in critical access rural hospitals. JAMA. 2011 Jul 6;306(1):45-52. doi: 10.1001/jama.2011.902. PMID 21730240
- [Derived] Levine DM, Desai MP, Findeisen SM, Blitzer SC, Brewster RCL, Grinman MN, Amrhein SC, Wicker M, Harrison SM, Dykes PC, Barthel MF, Lipsitz SR. Hospital-Level Care at Home for Adults Living in Rural Settings: A Randomized Clinical Trial. JAMA Netw Open. 2025 Dec 1;8(12):e2545712. doi: 10.1001/jamanetworkopen.2025.45712. PMID 41324962